CLINICAL TRIAL: NCT03114631
Title: Single-center Trial Evaluating the Safety and Efficacy of MUC-1/WT-1 Peptide or Tumor Lysate-pulsed Dendritic Cell Immunotherapy for the Patients With Pancreatic Cancer
Brief Title: Dendritic Cell Immunotherapy for the Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Principal Investigator, Andrei Y. Hancharou, Head of the Laboratory for Immunology and Cellular Biotechnology, The Republican Research and Practical Center for Epidemiology and Microbiology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRPCEM_DC1
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Dendritic Cells; Pancreatic Neoplasms
Keywords: dendritic cells, pancreatic cancer, immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dendritic cells lysate-pulsed group (Experimental): Patients treated according to clinical protocols plus autologous dendritic cells, pulsed with tumor lysate
  Interventions: Biological: Dendritic cells pulsed with tumor lysate
- Control group (No Intervention): Patients treated according to clinical protocols
- Dendritic cells peptide-pulsed group (Experimental): Patients treated according to clinical protocols plus autologous dendritic cells, pulsed with MUC-1/WT-1 peptides
  Interventions: Biological: Dendritic cells pulsed with MUC-1/WT-1 peptides

INTERVENTIONS:
Biological: Dendritic cells pulsed with tumor lysate
  Arms: Dendritic cells lysate-pulsed group
Biological: Dendritic cells pulsed with MUC-1/WT-1 peptides
  Arms: Dendritic cells peptide-pulsed group

SUMMARY:
The trial evaluates the safety and efficacy of MUC-1/WT-1 peptide and/or tumor lysate-pulsed dendritic cell Immunotherapy for the patients with pancreatic cancer

DETAILED DESCRIPTION:
The trial evaluates the safety and efficacy of dendritic cell Immunotherapy for the patients with pancreatic cancer. Dendritic cells are obtained from blood monocytes using standard protocol.

Two options for dendritic cell priming are used: MUC-1/WT-1 peptides for the patients with unresectable tumor and/or tumor lysates for the patients undergoing tumor resection.

The dendritic cells are them matured and injected subcutaneous (all patients) and intratumorally (when possible).

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed pancreatic cancer (adenocarcinoma);
* HLA-A2 expression by tumor cells;
* WT-1/MUC-1 expression by tumor cells.

Exclusion Criteria:

* refuse of patient to participate in the trial;
* pregnancy/lactation;
* intercurrent severe chronic diseases;
* HIV, Hepatites B/C;
* active tuberculosis;
* alcohol use disorder/drug addiction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with PR or CR at 1 year | 1 year
  1 year PR/CR
Number of Participants Who Survived at 1 Year | 1 year
  1 year overall survival

SECONDARY OUTCOMES:
Antigen-specific immune response | 1 year
  The increase of antigen-specific T-cells
Circulating tumor cells count | 1 year
  Decrease of EpCAM+CD45- circulating tumor cells count
Immune response | 1 year
  Decrease of T-regulatory cells
Number of Participants Who Survived at 2 Years | 2 years
  2 year overall survival
Number of Participants Who Survived at 3 Years or more | 3 years
  3 year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V. Prokharau, Prof., Study Director — Belarussian State Medical University, Minsk, Belarus; Andrei Y Hancharou, Dr., Study Director — The Republican Research and Practical Center for Epidemiology and Microbiology
Locations (1):
- Minsk City Clinical Oncologic Dispensary, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided